CLINICAL TRIAL: NCT00529763
Title: A Phase II Study to Determine the Activity of Dasatinib Administered Orally (PO) at a Dose of 100 mg Once Daily (QD) in Chronic Phase Chronic Myelogenous Leukemia (CML), at a Dose of 70 mg Twice Daily (BID) in Advanced Phase Chronic Myelogenous Leukemia (CML) Chinese Subjects Who Are Resistant to or Intolerant of Imatinib Mesylate (Gleevec®)
Brief Title: Dasatinib in Imatinib Resistant/Intolerant Chinese CML (Chronic and Advanced Phase) Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-160
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Results first posted 2011-04-05 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Leukemia
Keywords: Chronic Phase, Advanced Phase chronic myeloid leukemia; Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 70 mg BID (AD CML) or 100 mg QD (Chronic CML), once or twice daily dependent on disease stage, until subjects meet discontinuation (DC) criteria for study
  Other Names: Sprycel; BMS-354825

SUMMARY:
The primary objective of this study is to estimate the major cytogenetic response (MCyR) rate to Dasatinib in subjects with CP CML, complete and overall hematologic response (CHR and OHR) rate in subjects with AD CML or Ph+ ALL who have primary or acquired resistance to imatinib, or are intolerant of imatinib, when administered at 100 mg QD (Chronic CML) or 70mg BID (AP CML and Ph+ALL).

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Signed Written Informed Consent
* Men and women, ages 18 years of age or older
* Subjects with Chronic Phase (CP) or Advanced Disease (AD) chronic myeloid leukemia (CML)/Ph+ Acute Lymphoblastic Leukemia (Ph+ ALL)
* Subjects resistant/intolerant to imatinib
* Subjects presenting:

  1. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score 0-2
  2. Adequate hepatic function
  3. Adequate renal function
  4. Sodium, Potassium, Magnesium, Phosphorus, Calcium higher or equal than the lower limit of normal range

Exclusion Criteria:

* Women of child bearing potential who are not using adequate birth control
* Women who are pregnant or breastfeeding
* Subjects eligible for stem cell transplantation
* Serious uncontrolled medical disorder or active infection
* Uncontrolled or significant cardiovascular disease
* Concurrent incurable malignancy other than CML
* Subjects who received imatinib, interferon, cytarabine within 7 days or other antineoplastic agents other than hydroxyurea within 14 days before dasatinib, Dasatinib in the past
* History of significant bleeding unrelated to CML

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2007-11-17 (Actual); Primary Completion 2009-06-17 (Actual); Study Completion 2022-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- China (13):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution - 0004, Fuzhou, Fujian
  - Local Institution, Fuzhou, Fujian
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Nanjing, Jiangsu
  - Local Institution - 0008, Suzhou, Jiangsu
  - Local Institution, Suzhou, Jiangsu
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Chengdou, Sichuan
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Tianjin, Tianjin Municipality
  - Local Institution - 0009, Hangzhou, Zhejiang
  - Local Institution, Hangzhou, Zhejiang

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Advanced Disease CML - Accelerated Phase (AP): Participants with AP advanced disease CML who received prior treatment with imatinib mesylate and can no longer be treated with this drug due to primary or acquired resistance or intolerance. Dasatinib was administered orally at a dose of 70 mg BID. Participants were treated until progression of disease or intolerable toxicity as determined by the treating physician.
- Advanced Disease CML - Blast Phase/PH+ ALL: Participants with blast phase (BP) advanced disease CML or Philadelphia positive acute lymphoblastic leukemia (Ph+ALL) who received prior treatment with imatinib mesylate and can no longer be treated with this drug due to primary or acquired resistance or intolerance. Dasatinib was administered orally at a dose of 70 mg BID. Participants were treated until progression of disease or intolerable toxicity as determined by the treating physician.
- Chronic Phase (CP) CML: Participants with chronic phase (CP) CML who have received prior treatment with imatinib mesylate and can no longer be treated with this drug due to primary or acquired resistance or intolerance. Dasatinib was administered orally at a dose of 100 mg QD in patients with chronic phase CML. Participants were treated until progression of disease or intolerable toxicity as determined by the treating physician.
Period: Overall Study
Arm/Group | Advanced Disease CML - Accelerated Phase (AP) | Advanced Disease CML - Blast Phase/PH+ ALL | Chronic Phase (CP) CML
Started | 25 | 37 | 59
Completed (All participants who completed treatment were transitioned to the patient support program of Sprycel.) | 4 | 0 | 27
Not Completed | 21 | 37 | 32
Not completed — Adverse Event Unrelated to Study Drug | 1 | 5 | 3
Not completed — Death | 1 | 1 | 1
Not completed — Disease Progression | 10 | 16 | 11
Not completed — Lost to Follow-up | 1 | 2 | 3
Not completed — Stem Cell Transplant | 0 | 3 | 1
Not completed — Study Drug Toxicity | 3 | 6 | 4
Not completed — Participant Withdrew Consent | 2 | 3 | 4
Not completed — Other reasons | 2 | 0 | 2
Not completed — Participant request to discontinue treatment | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Advanced Disease CML - Accelerated Phase (AP) | Advanced Disease CML - Blast Phase/PH+ ALL | Chronic Phase (CP) CML | Total
Number analyzed (Participants) | 25 | 37 | 59 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (10.5) | 39.2 (13.4) | 42.8 (11.3) | 41.0 (11.9)
Age, Customized [Count of Participants; unit: Participants]
  <=21 years | 1 | 4 | 2 | 7
  Between 21 and 45 years | 18 | 23 | 33 | 74
  Between 46 and 65 years | 5 | 9 | 23 | 37
  Between 66 and 75 years | 1 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 23 | 42
  Male | 15 | 28 | 36 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 25 | 37 | 59 | 121
Region of Enrollment [Count of Participants; unit: Participants]
  China: China | 25 | 37 | 59 | 121
Eastern co-operative Oncology Group Performance Status (ECOG PS) [Number; unit: units on a scale] — ECOG PS, a 6-item scale to assess disease progression, daily functioning, and appropriate treatment and prognosis. Scale: 0-5, with 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Death. The inclusion criteria allowed only for scores of 0 to 2.
  units on a scale
    ECOG PS = 0 | 8 | 2 | 25 | 35
    ECOG PS = 1 | 16 | 29 | 33 | 78
    ECOG PS = 2 | 1 | 6 | 0 | 7
    Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Chronic Phase Chronic Myeloid Leukemia (CP - CML) Participants With Major Cytogenetic Response (MCyR)
Description: Major Cytogenetic Response (MCyR) is defined as Complete Cytogenetic Response (CCyR) or Partial Cytogenetic Response (PCyR).
  CCyR: 0% Ph-chromosome-positive cells in metaphase in bone marrow [BM] PCyR: 1-35% Ph-chromosome-positive cells in metaphase in [BM].
Time Frame: From first dose up to approximately 12 months of follow up after dasatinib treatment (data cut-off date: 18-Jun-2010)
Population: All treated participants with Chronic Phase Chronic Myeloid Leukemia (CP - CML). Data pre-specified to be collected in the Chronic Phase (CP) CML arm only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Chronic Phase (CP) CML
Number analyzed (Participants) | 59
Percentage of participants | 50.8 [37.5 to 64.1]

2. Primary Outcome: Percentage of Participants With Complete, Major, and Overall Hematologic Response (CHR, MaHR, & OHR) in Advanced Disease Chronic Myeloid Leukemia (AD CML) and Blast Phase CML/Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia (Ph+ ALL)
Description: Major hematologic response: (MaHR) = complete hematologic response (CHR) + no evidence of leukemia (NEL).
  CHR=white blood cells (WBC) ≤upper limit of normal (ULN); absolute neutrophil count (ANC) ≥1,000/mm3; platelets ≥100,000/mm3; no blasts/promyelocytes, <20% basophils & <5% myelocytes+metamyelocytes in peripheral blood (PB); BM blasts ≤5%; no extra-medullary involvement/hepatomegaly/splenomegaly.
  NEL=CHR except platelets ≥20,000/mm3 & <100,000/mm3; ANC >500/mm3 & <1,000/mm3.
  Overall hematologic response (OHR)=CHR+NEL+ return to chronic phase (RTC=<15% blasts in BM and PB; <30% blasts+promyelocytes in BM & PB; <20% basophils in PB; no extra-medullar disease other than spleen & liver)
Time Frame: From first dose up to approximately 12 months of follow up after dasatinib treatment (data cut-off date: 18-Jun-2010)
Population: All treated participants with Advanced Disease Chronic Myeloid Leukemia (CML). Data pre-specified to be collected in the Advanced Disease CML - AP and Blast Phase/PH+ ALL arms only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Advanced Disease CML - Accelerated Phase (AP) | Advanced Disease CML - Blast Phase/PH+ ALL
Number analyzed (Participants) | 25 | 37
Percentage of participants
  CHR | 52.0 [31.3 to 72.2] | 16.2 [6.2 to 32.0]
  MaHR | 84.0 [63.9 to 95.5] | 29.7 [15.9 to 47.0]
  OHR | 92.0 [74.0 to 99.0] | 35.1 [20.2 to 52.5]

3. Secondary Outcome: Percentage of Chronic Phase Chronic Myeloid Leukemia (CP - CML) Participants With Complete Hematologic Response (CHR)
Description: Complete Hematologic Response (CHR) is obtained when all the following criteria are met: WBC ≤ institutional ULN; platelets ≤ 450,000/mm3; ≤20% basophils in peripheral blood; no blasts or promyelocytes in PB cells; < 5% myelocytes plus metamyelocytes in PB cells; no extra-medullary involvement including no hepatomegaly or splenomegaly.
Time Frame: From first dose up to approximately 12 months of follow up after dasatinib treatment (data cut-off date: 18-Jun-2010)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Chronic Phase (CP) CML
Number analyzed (Participants) | 59
Percentage of participants | 91.5 [81.3 to 97.2]

4. Secondary Outcome: Time to Major Cytogenetic Response (MCyR) in Chronic Phase Chronic Myeloid Leukemia (CP - CML) Participants
Description: Time to MCyR is defined as the time from the first dosing date until day criteria were first met for CCyR or PCyR, whichever occurred first.
  Major Cytogenetic Response (MCyR) is defined as Complete Cytogenetic Response (CCyR: 0% Ph-chromosome-positive cells in metaphase in BM) or Partial Cytogenetic Response (PCyR: 1-35% Ph-chromosome-positive cells in metaphase in BM).
Time Frame: From first dose up to the day criteria were first met for CCyR or PCyR, whichever occurred first. (Up to approximately 12 months of follow up after dasatinib treatment [data cut-off date: 18-Jun-2010])
Population: All treated participants with Chronic Phase Chronic Myeloid Leukemia (CP - CML) with MCyR. Data pre-specified to be collected in the Chronic Phase (CP) CML arm only.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Chronic Phase (CP) CML
Number analyzed (Participants) | 30
Weeks | 12.1 [4.3 to 48.0]

5. Secondary Outcome: Duration of Major Cytogenetic Response (MCyR) in Chronic Phase Chronic Myeloid Leukemia (CP - CML) Participants
Description: The duration of time from when the first day all criteria are met for CCyR or PCyR until the date of progression or death. Participants who neither progress nor die will be censored on the date of their last cytogenetic assessment. The duration of MCyR will be estimated via the Kaplan-Meier product-limit method.
  Major Cytogenetic Response (MCyR) = Complete Cytogenetic Response (CCyR: 0% Ph-chromosome-positive cells in metaphase in BM) or Partial Cytogenetic Response (PCyR: 1-35% Ph-chromosome-positive cells in metaphase in BM).
Time Frame: From first dose until the date of progression or death. (Up to approximately 12 months of follow up after dasatinib treatment [data cut-off date: 18-Jun-2010])
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Chronic Phase (CP) CML
Number analyzed (Participants) | 30
Months | NA [NA to NA] — Insufficient number of participants with events

6. Secondary Outcome: Progression-free Survival Among CP CML Participants
Description: Progression-free survival is defined as the time from first dosing date until the time progressive disease (PD) is first documented. Participants who die without a reported prior progression will be considered to have progressed on the date of their death. Participants who do not progress nor die will be censored on the date of their last hematologic or cytogenetic assessment, whichever comes last. PFS will be analyzed via the Kaplan-Meier product-limit method.
  Participants were considered as having PD if they: achieved a hematologic response but subsequently no longer meet the criteria consistently on all assessment over a consecutive 2-week period after starting maximum dose; had no decrease from their baseline percent blasts in PB or BM on all assessments over a 4-week period, or had an increase by at least 50% in PB blast count (absolute) over a 2-week period after starting their maximum (individually-tolerated) dose.
Time Frame: From first dosing date until the time progressive disease (PD) is first documented. (Up to approximately 12 months of follow up after dasatinib treatment [data cut-off date: 18-Jun-2010])
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Chronic Phase (CP) CML
Number analyzed (Participants) | 59
Months | NA [NA to NA] — Insufficient number of participants with events

7. Secondary Outcome: Time to Complete and Major Hematologic Response (CHR and MaHR) in Advanced Disease Chronic Myeloid Leukemia (AD CML) and Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia Participants (Ph+ ALL)
Description: The time from first dose of Dasatinib until the first day CHR or MaHR criteria are met (for all confirmed responses). Time to CHR is computed only for participants whose best response is CHR. Major HR (MaHR) includes CHR or no evidence of leukemia (NEL).
  Major hematologic response: (MaHR) = complete hematologic response (CHR) + no evidence of leukemia (NEL).
  CHR=white blood cells (WBC) ≤upper limit of normal (ULN); absolute neutrophil count (ANC) ≥1,000/mm3; platelets ≥100,000/mm3; no blasts/promyelocytes, <20% basophils & <5% myelocytes+metamyelocytes in peripheral blood (PB); BM blasts ≤5%; no extra-medullary involvement/hepatomegaly/splenomegaly.
  NEL=CHR except platelets ≥20,000/mm3 & <100,000/mm3; ANC >500/mm3 & <1,000/mm3.
Time Frame: From first dose of Dasatinib until the first day CHR criteria are met (for all confirmed responses). (Up to approximately 12 months of follow up after dasatinib treatment [data cut-off date: 18-Jun-2010])
Population: All treated participants with Advanced Disease Chronic Myeloid Leukemia (CML) with CHR or MaHR. Data pre-specified to be collected in the Advanced Disease CML - AP and Blast Phase/PH+ ALL arms only.
Measure: Median (Full Range); unit: Weeks
Groups:
- Total: All treated Participants with Advanced Disease CML - Accelerated Phase (AP) and Blast Phase/PH+ ALL
Arm/Group | Advanced Disease CML - Accelerated Phase (AP) | Advanced Disease CML - Blast Phase/PH+ ALL | Total
Number analyzed (Participants) | 21 | 11 | 32
Weeks
  CHR: number analyzed (Participants) | 13 | 6 | 19
  CHR | 16.0 [11.7 to 52.1] | 12.1 [11.6 to 28.0] | 12.1 [11.6 to 52.1]
  MaHR | 12.1 [11.7 to 28.6] | 12.1 [11.6 to 24.0] | 12.1 [11.6 to 28.6]

8. Secondary Outcome: Duration of CHR Among AD CML and Ph+ ALL Participants
Description: Time from the first day all criteria are met for CHR until the date treatment is discontinued due to progressive disease (PD) or death. Participants who neither progress nor die will be censored on the date of their last assessment.
  CHR=white blood cells (WBC) ≤ upper limit of normal (ULN); absolute neutrophil count (ANC) ≥1,000/mm3; platelets ≥100,000/mm3; no blasts/promyelocytes, <20% basophils and <5% myelocytes+metamyelocytes in peripheral blood (PB); BM blasts ≤5%; no extra-medullary involvement/hepatomegaly/splenomegaly.
  PD = Hematologic response achieved but subsequently no longer meet the criteria consistently on all assessment over a 2-week period;, and no decrease from their baseline percent blasts in PB or BM on all assessments over a 4-week period or have an increase by at least 50% in PB blast count (absolute) over a 2-week period.
Time Frame: From first dose until the date of disease progression (PD) or death. (Up to approximately 12 months of follow up after dasatinib treatment [data cut-off date: 18-Jun-2010])
Population: All treated participants with Advanced Disease Chronic Myeloid Leukemia (CML) with CHR. Data pre-specified to be collected in the Advanced Disease CML - AP and Blast Phase/PH+ ALL arms only.
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Advanced Disease CML - Accelerated Phase (AP) | Advanced Disease CML - Blast Phase/PH+ ALL
Number analyzed (Participants) | 13 | 6
Months | NA [17.2 to NA] — Insufficient number of participants with events | NA [13.2 to NA] — Insufficient number of participants with events

9. Secondary Outcome: Duration of MaHR Among AD CML and Ph+ ALL Participants
Description: Time from the first day all criteria are met for CHR or NEL or MaHR until the date of progression or death. Participants who neither progress nor die will be censored on the date of their last assessment.
  MAHR = CHR or no evidence of leukemia (NEL). CHR=white blood cells (WBC) ≤ upper limit of normal (ULN); absolute neutrophil count (ANC) ≥1,000/mm3; platelets ≥100,000/mm3; no blasts/promyelocytes, <20% basophils and <5% myelocytes+metamyelocytes in peripheral blood (PB); BM blasts ≤5%; no extra-medullary involvement/hepatomegaly/splenomegaly.
  NEL=CHR except platelets ≥20,000/mm3 and <100,000/mm3; ANC >500/mm3 and <1,000/mm3.
  Progressive disease (PD) = Hematologic response achieved but subsequently no longer meet the criteria consistently on all assessment over a 2-week period;, and no decrease from their baseline percent blasts in PB or BM on all assessments over a 4-week period or have an increase by at least 50% in PB blast count (absolute) over a 2-week period.
Time Frame: as for outcome 8
Population: All treated participants with Advanced Disease Chronic Myeloid Leukemia (CML) with CHR or NEL or MiHR. Data pre-specified to be collected in the Advanced Disease CML - AP and Blast Phase/PH+ ALL arms only.
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Advanced Disease CML - Accelerated Phase (AP) | Advanced Disease CML - Blast Phase/PH+ ALL
Number analyzed (Participants) | 21 | 11
Months | NA [22.9 to NA] — Insufficient number of participants with events | 11.2 [2.8 to NA] — Insufficient number of participants with events

10. Secondary Outcome: Progression-free Survival Among AD CML and Ph+ ALL Participants
Description: Progression-free survival is defined as the time from first dosing date until the time progressive disease (PD) is first documented. Participants who die without a reported prior progression will be considered to have progressed on the date of their death. Participants who do not progress nor die will be censored on the date of their last hematologic or cytogenetic assessment whichever comes last. PFS will be analyzed via the Kaplan-Meier product-limit method.
  Progressive disease (PD) = Hematologic response achieved but subsequently no longer meet the criteria consistently on all assessment over a 2-week period;, and no decrease from their baseline percent blasts in PB or BM on all assessments over a 4-week period or have an increase by at least 50% in PB blast count (absolute) over a 2-week period.
Time Frame: From first dose until the time progressive disease (PD) is first documented. (Up to approximately 12 months of follow up after dasatinib treatment [data cut-off date: 18-Jun-2010])
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Advanced Disease CML - Accelerated Phase (AP) | Advanced Disease CML - Blast Phase/PH+ ALL
Number analyzed (Participants) | 25 | 37
Months | 25.7 [20.3 to NA] — Insufficient number of participants with events | 4.3 [2.6 to 7.4]

11. Secondary Outcome: Deaths, Serious Adverse Events (SAEs), Adverse Events (AEs), and Drug-related Fluid Retention AEs of Special Interest
Description: AEs and SAEs considered possibly, probably, or certainly related to study treatment, graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 (Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death).SAE= any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization/prolongation of existing hospitalization, results in persistent/significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: From first dose to 30 days after last dose. (Up to approximately 161 months)
Population: All treated participants
Measure: Number; unit: Participants
Arm/Group | Chronic Phase (CP) CML | Advanced Disease CML - Accelerated Phase (AP) | Advanced Disease CML - Blast Phase/PH+ ALL
Number analyzed (Participants) | 59 | 25 | 37
Participants
  Deaths | 4 | 4 | 13
  All-Causality SAEs | 18 | 13 | 24
  Drug-Related SAEs | 10 | 8 | 11
  All-Causality AEs Leading to Discontinuation | 10 | 9 | 19
  Drug-Related AEs leading to Discontinuation | 6 | 3 | 6
  All AEs | 52 | 25 | 33
  Drug-Related AEs | 46 | 21 | 30
  Drug-Related Gr3/4 AEs | 14 | 16 | 21
  Drug-related Fluid Retention-related AEs (FR AE) - Ascites | 2 | 0 | 0
  Drug-related FR AE - Pleural Effusion | 16 | 13 | 10
  Drug-related FR AE - Pulmonary Hypertension | 5 | 3 | 0
  Drug-related FR AE - Oedema Peripheral | 2 | 1 | 0
  Drug-related FR AE - Pericardial Effusion | 2 | 5 | 2
  Drug-related FR AE - Oedema | 0 | 2 | 1

12. Secondary Outcome: Mean Dasatinib Plasma Concentrations
Description: Mean dasatinib plasma concentrations following 70 mg BID dose in AD CML or Ph+ ALL participants and following 100 mg QD dose in CP CML participants
Time Frame: Day 1 (0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours postdose), Days 6 and 7 (0 hours postdose), Day 8 (0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12 hours postdose),
Population: All treated participants with evaluable PK data. Data collection pre-specified by treatment dosage.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 70 mg BID: Participants with AP CML or Ph+ ALL treated with 70 mg dasatinib BID
- 100 mg QD: Participants with CP CML treated with dasatinib 100 mg QD
Arm/Group | 70 mg BID | 100 mg QD
Number analyzed (Participants) | 11 | 11
ng/mL
  Day 1: 0.5 hours postdose: number analyzed (Participants) | 10 | 10
  Day 1: 0.5 hours postdose | 56.74 (59.71) | 133.18 (116.06)
  Day 1 : 1 hour postdose | 54.57 (44.06) | 130.86 (81.56)
  Day 1 : 2 hours postdose | 29.50 (24.87) | 100.69 (60.37)
  Day 1 : 3 hours postdose | 16.65 (12.23) | 64.90 (31.15)
  Day 1 : 4 hours postdose | 12.02 (7.95) | 38.18 (16.48)
  Day 1 : 5 hours postdose | 8.53 (4.51) | 26.33 (11.83)
  Day 1 : 6 hours postdose | 7.37 (4.89) | 20.71 (9.91)
  Day 1 : 8 hours postdose: number analyzed (Participants) | 10 | 11
  Day 1 : 8 hours postdose | 4.48 (2.21) | 14.00 (7.25)
  Day 1 : 12 hours postdose: number analyzed (Participants) | 8 | 11
  Day 1 : 12 hours postdose | 2.42 (0.93) | 6.57 (3.82)
  Day 1 : 24 hours postdose: number analyzed (Participants) | 2 | 7
  Day 1 : 24 hours postdose | 1.07 (0.08) | 2.59 (1.43)
  Day 6: 0 hours postdose: number analyzed (Participants) | 11 | 8
  Day 6: 0 hours postdose | 8.93 (4.24) | 3.15 (3.57)
  Day 7: 0 hours postdose: number analyzed (Participants) | 11 | 9
  Day 7: 0 hours postdose | 8.77 (4.40) | 3.02 (2.03)
  Day 8: 0 hours postdose: number analyzed (Participants) | 11 | 10
  Day 8: 0 hours postdose | 8.22 (3.41) | 2.75 (1.58)
  Day 8: 0.5 hours postdose | 48.74 (56.24) | 102.69 (92.00)
  Day 8: 1 hours postdose | 52.55 (39.79) | 168.51 (112.14)
  Day 8: 2 hours postdose | 44.32 (31.31) | 102.05 (69.80)
  Day 8: 3 hours postdose | 31.64 (19.93) | 71.23 (34.29)
  Day 8: 4 hours postdose | 18.33 (9.66) | 45.17 (20.04)
  Day 8: 5 hours postdose | 13.74 (6.36) | 31.16 (13.47)
  Day 8: 6 hours postdose | 10.91 (5.09) | 23.62 (12.13)
  Day 8: 8 hours postdose | 7.23 (3.28) | 15.41 (8.04)
  Day 8: 12 hours postdose: number analyzed (Participants) | 10 | 11
  Day 8: 12 hours postdose | 3.96 (1.62) | 7.55 (3.90)

13. Secondary Outcome: Mean Maximum Concentration (Cmax) of Dasatinib Following 70 mg BID and 100 QD Dose Administration
Description: Cmax=maximum observed plasma concentration of dasatinib
Time Frame: Day 1 (0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours postdose), Day 8 (0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12 hours postdose)
Population: All treated participants with evaluable PK data. Data collection pre-specified by treatment dosage.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 70 mg BID | 100 mg QD
Number analyzed (Participants) | 11 | 11
ng/mL
  Day 1 | 71.01 (54.705) | 170.53 (99.245)
  Day 8 | 71.54 (51.908) | 181.79 (94.689)

14. Secondary Outcome: Mean (Tmax) and (T-Half) of Dasatinib Following 70 mg BID and 100 QD Dose Administration
Description: Tmax=time of maximum observed plasma concentration. T-Half=plasma half-life.
Time Frame: Day 1 (0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours postdose), Day 8 (0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12 hours postdose)
Population: All treated participants with evaluable PK data. Data collection pre-specified by treatment dosage.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 70 mg BID | 100 mg QD
Number analyzed (Participants) | 11 | 11
hours
  Tmax: Day 1 | 1.17 (1.348) | 1.50 (0.947)
  Tmax: Day 8 | 1.62 (0.896) | 1.23 (0.684)
  T-Half: Day 1 | 4.35 (2.445) | 4.78 (1.679)
  T-Half: Day 8 | 4.80 (1.660) | 5.71 (1.012)

15. Secondary Outcome: Mean (AUC[0-T]), (AUC[INF]), and (AUC[TAU])of Dasatinib Following 70 mg BID and 100 QD Dose Administration
Description: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration AUC(0-T)for dasatinib. AUC(INF)=area under the plasma concentration-time curve from time zero extrapolated to infinite time. AUC(TAU)=area under the plasma concentration-time curve for a dosing interval
Time Frame: Day 1 (0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours postdose), Day 8 (0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12 hours postdose)
Population: All treated participants with evaluable PK data. Data collection pre-specified by treatment dosage.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | 70 mg BID | 100 mg QD
Number analyzed (Participants) | 11 | 11
ng*h/mL
  AUC(0-T): Day 1 | 161.30 (104.266) | 505.73 (214.365)
  AUC(0-T): Day 8 | 214.60 (102.616) | 567.30 (286.851)
  AUC(INF): Day 1 | 174.26 (105.824) | 526.33 (216.351)
  AUC(INF): Day 8 | 247.10 (103.802) | 588.52 (293.512)
  AUC(TAU): Day 1 | 163.56 (103.573) | 511.07 (211.781)
  AUC(TAU): Day 8 | 218.05 (104.156) | 568.85 (285.532)

16. Secondary Outcome: Mean Oral Clearance (CLo) of Dasatinib Following 70 mg BID and 100 QD Dose Administration
Time Frame: Day 1 (0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours postdose), Day 8 (0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12 hours postdose)
Population: All treated participants with evaluable PK data. Data collection pre-specified by treatment dosage.
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | 70 mg BID | 100 mg QD
Number analyzed (Participants) | 11 | 11
mL/h
  Day 1 | 564.97 (318.555) | 221.84 (99.003)
  Day 8 | 441.08 (307.574) | 211.09 (88.089)

17. Secondary Outcome: Mean Apparent Volume of Distribution (Vz/F) of Dasatinib Following 70 mg BID and 100 QD Dose Administration
Time Frame: Day 1 (0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours postdose), Day 8 (0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12 hours postdose)
Population: All treated participants with evaluable PK data. Data collection pre-specified by treatment dosage.
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | 70 mg BID | 100 mg QD
Number analyzed (Participants) | 11 | 11
mL/h
  Day 1 | 3785.78 (3034.812) | 1454.71 (604.728)
  Day 8 | 3446.74 (3196.014) | 1719.14 (730.345)

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their study completion (up to approximately 173 months). AE and SAEs were collected form first dose to 30 days post last dose (up to approximately 161 months) .
Arm/Group | Advanced Disease CML - Accelerated Phase (AP) | Advanced Disease CML - Blast Phase/PH+ ALL | Chronic Phase (CP) CML
All-Cause Mortality (participants affected / at risk) | 5/25 | 16/37 | 5/59
Serious Adverse Events (participants affected / at risk) | 13/25 | 24/37 | 18/59
Other Adverse Events (participants affected / at risk) | 24/25 | 30/37 | 50/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Advanced Disease CML - Accelerated Phase (AP) (N=25) | Advanced Disease CML - Blast Phase/PH+ ALL (N=37) | Chronic Phase (CP) CML (N=59)
Bone marrow necrosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 1
Oedema (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0
Sudden death (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Anal infection (Infections and infestations) | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 6 | 1
Respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Peripheral nerve injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 7 | 1
Chronic myeloid leukaemia transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Central nervous system haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Intracranial haematoma (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Allogenic bone marrow transplantation therapy (Surgical and medical procedures) | 0 | 2 | 0
Bone marrow transplant (Surgical and medical procedures) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Advanced Disease CML - Accelerated Phase (AP) (N=25) | Advanced Disease CML - Blast Phase/PH+ ALL (N=37) | Chronic Phase (CP) CML (N=59)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 10
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 7 | 4 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 4 | 9
Palpitations (Cardiac disorders) | 0 | 0 | 3
Pericardial effusion (Cardiac disorders) | 5 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 3
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 4 | 6
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 3
Chest discomfort (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 6
Pyrexia (General disorders) | 4 | 8 | 7
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 3 | 0
Infection (Infections and infestations) | 4 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 6
Oral infection (Infections and infestations) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 8 | 7 | 6
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 6
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 4
Headache (Nervous system disorders) | 4 | 2 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 9 | 14
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Hypertension (Vascular disorders) | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.